CLINICAL TRIAL: NCT07072897
Title: Restrictive Versus Liberal Fluid Therapy in Patients Undergoing Pancreaticoduodenectomy: A Prospective Randomized Controlled Study
Brief Title: A Study Comparing Restrictive and Liberal Fluid Therapy During Pancreatecoduodenectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Romi Dahal, principal investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nepalhealthresearchcouncil2379
Record Dates: First submitted 2025-06-22; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer, Resected; Whipple Procedure
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- restrictive fluid therapy (Experimental): Restrictive fluid therapy given as bolus of 5ml/kg/hr and the same amount of fluid (5ml/kg/hr) was continued as intraoperative requirement till the end of surgery. Fluid in the restrictive group given postoperatively at the rate of 1ml/kg/hr. This fluid to be given till the 24 hours of the start of surgery which was the study period for this trial. Treating physician was more inclined towards the use of noradrenaline for the maintenance of BP if the urine output was adequate (>0.5ml/kg/hr).
  Interventions: Other: Fluid bolus administration
- liberal fluid therapy (Active Comparator): In the liberal fluid therapy arm, intraoperatively the patients receive a fixed dose of fluid with a bolus of 10ml/kg/hr followed by 10ml/kg/hr till the completion of surgery. The patients receive fluid at the rate of 1.5ml/kg/hr in the postoperative period until 24 hours of the start of surgery.
  Fluid boluses of 250ml each to be given anytime during the study period to overcome hypotension or oliguria (<0.5ml/kg/hr) if felt necessary by the physician.
  Furosemide 10mg given intravenously anytime if the clinician was suspicious of fluid overload during the study period.
  Interventions: Other: Frusemide was given when required

INTERVENTIONS:
Other: Fluid bolus administration — fluid boluses 250 ml were given when required
  Arms: restrictive fluid therapy
Other: Frusemide was given when required — fluid is given in a fixed regimen
  Arms: liberal fluid therapy

SUMMARY:
ancreaticoduodenectomy (also known as PD or the Whipple procedure) is a major surgery often done for conditions like pancreatic cancer. Over the past few decades, doctors around the world have greatly improved surgical techniques, reducing the risk of death after PD from about 24% in the 1980s to less than 2% today in good volume hospitals.

However, even though fewer patients are dying from the surgery, many still face complications after surgery, such as infections, delayed healing, or other problems called as morbidities. These problems can affect 17% to 50% of patients.

One important factor that may affect recovery is fluid management - the amount of fluids patients receive around the time of surgery.

Traditionally, surgeons gave large amounts of fluid during and after surgery, thinking it helped keep blood pressure and urine output stable. This approach is called liberal fluid therapy. But giving too much fluid can cause swelling, weight gain, and slower recovery.

A newer method, called restrictive fluid therapy, gives smaller, more controlled amounts of fluid to avoid these problems. This approach is new and has shown good results in some studies however the exact role is yet unclear.

At our hospital, we usually use liberal fluid therapy and give fluids based on the treating physician, using these fluids or restricting them as per the treating physician's choice.

So, the study compares these two fluid strategies in patients having PD. Our goal is to find out whether using less fluid (restrictive therapy) could help reduce complications and improve patient outcomes when compared to using more liberal fluids.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent PD at TUTH during the research duration.
* All patients above 18 years.

Exclusion Criteria:

* Those not willing to participate in the study.
* All patients with age ≥ 75 years.
* Patients with Chronic renal failure.
* Patients with major Cardiac illness.
* Patients who died within 24 hours of surgery.
* Failure to comply with the regimen due to any reason.
* Those who underwent palliative procedure instead of planned PD.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
postoperative complications CD≥ IIIb | 1 month
  CD IIIb and more were chosen as major complications as major morbidity occurs when the patient is taken to operating room or ICU to manage these complications.

SECONDARY OUTCOMES:
other complications | 1 month
  Other complications were procedure specific complications like POPF,DGE and other complications that can occur after pancreaticoduodenectomy like Pneumonia, SSI

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
IPD including demographic data and outcomes will be shared with qualified researchers upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 mth to 5 yeas of publication
Access Criteria: Access will be granted upon review and approval by the principal investigator and with a signed data use agreement. Requests should be sent to srgeon1@gmail.com

REFERENCES:
- [Background] Myles P, Bellomo R, Corcoran T, Forbes A, Wallace S, Peyton P, Christophi C, Story D, Leslie K, Serpell J, McGuinness S, Parke R; Australian and New Zealand College of Anaesthetists Clinical Trials Network, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus liberal fluid therapy in major abdominal surgery (RELIEF): rationale and design for a multicentre randomised trial. BMJ Open. 2017 Mar 3;7(3):e015358. doi: 10.1136/bmjopen-2016-015358. PMID 28259855
- See also: Peer-reviewed publication related to the study rationale and background — https://pubmed.ncbi.nlm.nih.gov/36688507